CLINICAL TRIAL: NCT04396652
Title: Comparison of Adductor Canal Block, Peri-articular Injection or Infiltration Between Popliteal Artery and Posterior Knee Capsule (IPACK) With Adductor Canal Block in Total Knee Arthroplasty.
Brief Title: Peri-articular Injection and (IPACK) With Adductor Canal Block in Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Shebl Abdelghany, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 33748/3/20; Tanta University (Other: Faculty of Medicine, Tanta University)
Record Dates: First submitted 2020-05-05; First posted 2020-05-20 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain; Regional Anesthesia
Keywords: peri-articular injection; adductor canal block; IPACK; Total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: * The patients will be blind through the use of closed sealed envelops.
  * The measurement will be collected by anesthesia nurse not participating in the study and blinded to its group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adductor canal block (ACB) group (Experimental): Patients will receive ACB under ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.25% Levobupivacaine will be injected in the canal
  Interventions: Procedure: Adductor canal block (ACB) group
- Peri-articular injection group (Experimental): Patients in group II will receive intraoperative peri-articular (cocktail) injection and will be performed by a single surgeon.
  A periarticular cocktail injection consisting of 90 mL of normal saline, 17.5 mL of 0.5% levobupivacaine, 2 mL of ketorolac (30 mg), and 0.5mg (0.5mL) of adrenaline, The total volume of the cocktail will be 110 mL
  Interventions: Procedure: Peri-articular injection group
- Adductor canal block and IPACK block group (Experimental): Patients will receive ACB under ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.25% Levobupivacaine will be injected in the canal IPACK block in which The ultrasound probe will be positioned in the popliteal crease, and needle will be inserted into the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur and 15 ml of 0.25% Levobupivacaine will be injected
  Interventions: Procedure: Adductor canal block and IPACK block group

INTERVENTIONS:
Procedure: Adductor canal block (ACB) group — Patients will receive ACB under ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.25% Levobupivacaine will be injected in the canal
  Arms: Adductor canal block (ACB) group
Procedure: Peri-articular injection group — Patients in group II will receive intraoperative peri-articular (cocktail) injection and will be performed by a single surgeon.
  A periarticular cocktail injection consisting of 90 mL of normal saline, 17.5 mL of 0.5% levobupivacaine, 2 mL of ketorolac (30 mg), and 0.5mg (0.5mL) of adrenaline, The total volume of the cocktail will be 110 mL
  Arms: Peri-articular injection group
Procedure: Adductor canal block and IPACK block group — Patients will receive ACB under ultrasound guidance in which the adductor canal was identified beneath the sartorius muscle and 20 ml of 0.25% Levobupivacaine will be injected in the canal IPACK block in which The ultrasound probe will be positioned in the popliteal crease, and needle will be inserted into the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur and 15 ml of 0.25% Levobupivacaine will be injected
  Arms: Adductor canal block and IPACK block group

SUMMARY:
This is a prospective randomized double blind controlled study to evaluate the post-operative analgesic effect of adductor canal block (ACB) or peri-articular injection (PAIs) compared to combined adductor canal block and infiltration of the interspace between popliteal artery and the capsule of posterior knee block ( IPACK) in patient undergoing total knee arthroplasty

DETAILED DESCRIPTION:
This prospective randomized study will be carried out in Tanta University Hospitals in Anesthesia Department for one year after approval from ethical committee of faculty of medicine of Tanta university. After approval from institutional ethics committee, an informed consent will be taken from each patient. All data of the patients will be confidential with secret codes and private file for each patient, all given data will be used for the current medical research only. Any unexpected risks encountered during the course of the research will be cleared to the participants as well as to the Ethical Committee on time. Every patient will receive an explanation to the purpose of the study and every patient will have a secret code number to ensure privacy to participants and confidentiality of data.

Inclusion criteria:

Adult patients with severe osteoarthritis , ASA class I, II and III and scheduled for elective Total knee arthroplasty will be enrolled in the study.

Exclusion criteria:

* Patient who refuse the regional anesthesia technique.
* History of allergy to local anesthetics.
* Local infection at the site of the block.
* Patients with bleeding and coagulation disorders.
* Patient with Advanced renal, hepatic and cardiac diseases.
* Preexisting lower extremity neurological abnormality, or neuropathy and difficulties in comprehending (NRS).

Grouping and Allocation:

60 patients will be enrolled in this study in each group, Patients will be randomly classified into three equal groups (20 patients each).

Randomization will be done by computer generated numbers into:

Group (I): 20 patients will receive adductor canal block alone. Group (II): 20 Patients will receive peri-articular injection alone. Group (III): 20 patients will receive adductor canal block (ACB) and infiltration of the interspace between popliteal artery and the capsule of posterior knee block (IPACK).

Anesthetic technique:

Preoperative assessment will be done by:

History talking, clinical examination, routine laboratory investigations including CBC, coagulation profile, random blood sugar, liver and renal function tests. During the pre-anesthetic assessment, all patients will be familiarized with Numeric Rating Scale (NRS) score. On entering the operating room, intravenous line (IV) will be inserted, routine monitoring of heart rate by ECG, noninvasive blood pressure (NIBP), pulse oximetry will be done. All patients will receive spinal anesthesia with 3 ml 0.5% (15 mg) hyperbaric bupivacaine plus 25 μgm fentanyl at the L3/4 interspaces and the study of regional anesthetic technique will be performed postoperatively according to each group. All patients will receive postoperative analgesic regimen which is paracetamol 1gm intravenously every 8 hours and ketorolac 30mg every12 hours. Rescue analgesia in the form of 0.05 mg/kg of morphine IV will be administrated when the Numeric Rating Score (NRS) exceeding 3. The morphine dose will be repeated whenever indicated considering the total dose in the first 24 hours never exceeding 20 mg.

Measurements:

1. Demographic data (age, gender, weight, ASA classification).
2. Post-operative pain will be assessed by Numeric Rating Scale (NRS) from 0 to 10 at 0,2,4,6 then every 6h for 24 hours and in the second and third postoperative days at rest and during Physiotherapy.
3. Postoperative analgesia, which will be assessed by total analgesic consumption, and time till administration of first rescue analgesia will be recorded.
4. Effect on Motor function: by recording the mean time taken to achieve 90o active knee flexion each day till the third postoperative day.
5. Adverse effects: hypotension, Bradycardia, infection, hematoma and local anesthetic toxicity will be observed and treated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe osteoarthritis , ASA class I, II and III and scheduled for elective Total knee arthroplasty

Exclusion Criteria:

* Patient who refuse the regional anesthesia technique.
* History of allergy to local anesthetics.
* Local infection at the site of the block.
* Patients with bleeding and coagulation disorders.
* Patient with Advanced renal, hepatic and cardiac diseases.
* Preexisting lower extremity neurological abnormality, or neuropathy and difficulties in comprehending (NRS)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | After the resolution of the effect of spinal anesthesia for 72 hours postoperative
  Post-operative pain will be assessed at rest and during physiotherapy by Numeric Rating Scale from (0-10) '0' representing "no pain" to '10' representing "worst pain imaginable"

SECONDARY OUTCOMES:
Postoperative analgesia | First 24 hours postoperatively
  Total analgesic consumption will be recorded
Duration of the block | First 24 hours postoperatively
  Time till administration of first rescue analgesia will be recorded
Effect on Motor function | Each day till the third postoperative day
  By recording the mean time taken to achieve 90o active knee flexion

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Abdelghany, Lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers